CLINICAL TRIAL: NCT02369133
Title: Preemptive Analgesia With Intravenous Paracetamol for Post-cesarean Section Pain Control : A Randomized Controlled Trial
Brief Title: Preemptive Analgesia With Intravenous Paracetamol for Post-cesarean Section Pain Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ozlem Ozmete, Medical Doctor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA 13-180
Record Dates: First submitted 2015-02-17; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Cesarean Section; Dehiscence
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Paracetamol (Group P), (Active Comparator): Drugs were given intravenously by a nurse unaware of the study 15 min before surgery. Patients in group P (n = 30) received 1 g iv paracetamol
  Interventions: Drug: paracetamol
- Group Saline (Group S) (Placebo Comparator): Drugs were given intravenously by a nurse unaware of the study 15 min before surgery. Patients in group S (n = 30) received 100 ml iv %0,9 saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: paracetamol — Drugs were given intravenously by a nurse unaware of the study 15 min before surgery. Patients in group P (n = 30) received 1 g iv paracetamol, patients in group S (n = 30) received 100 ml iv %0.9 NaCl
  Arms: Group Paracetamol (Group P),
Drug: Placebo
  Arms: Group Saline (Group S)

SUMMARY:
The investigators designed a prospective randomized study to investigate the efficacy of intravenous (IV) preemptive paracetamol on postoperative pain scores, patient satisfaction, total morfin consumption and the incidence of morfin-related side effects in patients undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 20-40 years,
* ASA physical status 1-2 who underwent elective cesarean surgery during general anesthesia were included in the study

Exclusion Criteria:

* A history of allergy to any of the study medications (opiod, general anesthetic agents or paracetamol),
* history of opioid or paracetamol use,
* hepatic or renal failure,
* any psychological disorders,
* complications during cesarean section and unable to use PCIA device were excluded from the study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores measured by visual analog scale (VAS) | Postoperative 24 hours